CLINICAL TRIAL: NCT03652922
Title: Propranolol Reactivation Mismatch (PRM) Treatment for PTSD: A Pilot Study
Brief Title: Propranolol Reactivation Mismatch (PRM) Treatment for PTSD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Roger K. Pitman, MD, Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018P001517
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propranolol (Experimental)
  Interventions: Drug: Reactivation Mismatch
- Placebo (Placebo Comparator)
  Interventions: Drug: Reactivation Mismatch

INTERVENTIONS:
Drug: Reactivation Mismatch — Ninety minutes prior to each of six weekly traumatic memory reactivation sessions, the subject will be given 0.67 mg/kg of short-acting propranolol (or placebo), rounded up to the nearest 10 mg (minimum 40 mg) and 1 mg/kg of oral long-acting propranolol or placebo (minimum 60 mg). rounded so as to achieve a dose of 60, 80, 120, or 160 mg. The subject will then read a narrative of their personal traumatic event aloud. During each weekly reading, a simple, different "mismatch" condition will be created by having the subject do such things as whisper the narrative, skip over every word that contains the letter "e," pronounce the narrative in a different accent, or alter the tense and/or person of the narrative.

SUMMARY:
The aim of the proposed work is to gather pilot data from an attempt to enhance the ability of propranolol reactivation (PR) to improve PTSD symptoms by incorporating into the design a mismatch (PRM) between what is expected and what occurs while a subject reads a narrative of the traumatic event that caused their PTSD under the influence of the ß-adrenergic blocking drug propranolol. It is hypothesized that a series of PRM treatments will produce superior symptomatic decreases compared to what the investigators have found in prior, published studies using PR without mismatch.

Under certain circumstances, retrieval (reactivation) of a traumatic memory returns it to a deconsolidated state from which it must be reconsolidated if it is to persist. Concomitant administration of the ß-adrenergic blocker weakens a deconsolidated traumatic memory and reduces PTSD symptoms, presumably through blockade of reconsolidation. It has recently been discovered that in order for deconsolidation to occur, there must be a mismatch between what is expected and what actually occurs. Altering the context in which a traumatic memory is retrieved putatively represents a deconsolidation-promoting mismatch. Experimentally increasing mismatch by manipulating context may make propranolol more effective in the treatment of PTSD.

The design is a single-blind, placebo-controlled, randomized PRM clinical trial by Partners researchers in 11 convenience pilot subjects between ages 18 and 65 with active PTSD, using a 10:1 propranolol:placebo randomization schedule. This two-month study will have the following components: Pre-treatment psychometric evaluation; Treatment consisting of six weekly PRM sessions with propranolol, or placebo; Post-treatment psychometric evaluation; Six-month follow-up psychometric evaluation. The Clinician-Administered PTSD Scale (CAPS) and PTSD Checklist (PCL) will be administered at pre- and post-treatment and at follow-up. The Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders-fifth edition (DSM-5) will also be administered at the pre-treatment evaluation. The PCL will also be administered prior to each weekly treatment session.

Pilot data analysis will consist of calculation of percent improvements and effect sizes in CAPS-5 and PCL-5 scores; observational comparisons with results obtained without mismatch in prior published studies; informal statistical comparisons via t-tests; and calculation of effect sizes for power analysis for a subsequent definitive study, if indicated.

ELIGIBILITY:
Inclusion Criteria

• Convenience sample of pilot subjects between ages 18 and 65 with active PTSD

Exclusion Criteria

* Age <18 or >65;
* Basal systolic blood pressure <100 mm Hg or heart rate <55 beats per minute;
* Medical condition that contraindicates the administration of propranolol, e.g., history of congestive heart failure, heart block, insulin-requiring diabetes, chronic bronchitis, emphysema, or asthma. With regard to asthma, because many persons who say they have had an asthma attack, especially as a child, may only have had hay fever, another allergy, or another non-asthmatic episode, a blanket exclusion criterion may be overly restrictive. Therefore, asthma attacks will only be exclusionary if they a.) occurred within the past ten years, b.) occurred at any time in life if induced by a β-blocker, or c.) are currently being treated, regardless of the date of last occurrence;
* Previous adverse reaction to, or non-compliance with, a β-blocker
* Current use of medication that may involve potentially dangerous interactions with propranolol, including, other β-adrenergic blockers, antiarrhythmics, calcium channel blockers and benzodiazepines. Subjects taking an α-1-adrenergic antagonist (e.g., prazosin) or an α -1-adrenergic agonist (e.g., clonidine) will be asked to refrain from taking this medication on the day of a study medication visit. Note: Possible inhibition of CYP2D6 isoenzyme-dependent reactions will not be of concern in this study, because propranolol will only be administered once a week for six weeks;
* Presence of drugs of abuse, including opiates, marijuana, cocaine, or amphetamines, as determined by saliva or urine testing;
* Pregnancy or breast feeding. Women of childbearing age will have a pregnancy test prior to being administered study medication at study week 0, and again at study week 7, following study medication discontinuation;
* Current PTSD from a traumatic event other than the event being treated, or another contraindicating psychiatric condition, e.g., current psychotic, bipolar, melancholic, or active substance dependence or abuse disorder;
* Initiation of, or change in, psychotropic medication within the previous two months. For subjects receiving stable doses of pharmacotherapy, they and their providers will be asked not to change the regimen during the proposed two-month study (excluding the 6-month follow-up) except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis with regard to retaining the subject or terminating participation
* Current participation in any psychotherapy (other than supportive). Subjects will be asked not to initiate new psychotherapy during the proposed two-month study (excluding the 6-month follow-up) except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis with regard to retaining the subject or terminating participation;
* Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation;
* Subject candidate does not understand English. This exclusion criterion is necessary because the procedures require a subtle dialogue with solely English-speaking investigators, which translation cannot accomplish. There is a need for rapid communication with English-speaking investigators in case of an adverse drug effect.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) Change Score | Change from Baseline at Week 0 to Post-Treatment at Week 7
  The PCL-5 is a published, validated, 20-item questionnaire, corresponding to the DSM-5 symptom criteria for PTSD. The self-report rating scale is 0-4 for each symptom. Possible scores range from 0 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Pitman, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Undecided